CLINICAL TRIAL: NCT01544621
Title: Escape Smoke Project: Non-Intervention Multicenter Study On the Real-Life Effectiveness of Smoking Cessation in General Practice in Denmark
Brief Title: Escape Smoke Project: Non-Intervention Non-Drug Multicenter Study on the Real-life Effectiveness of Smoking Cessation in General Practice in Denmark
Acronym: ESCAPE SMOKE
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Collaborators: Technical University of Denmark (DTU) (Unknown)
Responsible Party: Sponsor
Other Study IDs: A3051150
Record Dates: First submitted 2012-02-29; First posted 2012-03-06 (Estimated); Last update posted 2013-05-21 (Estimated); Status verified 2013-05

CONDITIONS: Smoking Cessation
Keywords: Real life smoking cessation. NON-drug NON-intervention study
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Successful quitters Sustained smokers: Successful quitters
  Interventions: Other: Smoking cessation

INTERVENTIONS:
Other: Smoking cessation — Smoking cessation

SUMMARY:
Real life smoking cessation rates after 24 weeks non-intervention design. Approximately 40 General Practice (GP) centers with 800 smokers will participate.

DETAILED DESCRIPTION:
Active smokers who wish to quit seen at in primary care practices

ELIGIBILITY:
Inclusion Criteria:

* Smoking males or females aged 18 years or older.
* Subjects being motivated for and willing to quit smoking.
* Ability to read and understand Danish.

Exclusion Criteria:

* Not smoking.
* Aged below 18 years.
* Lack of motivation and willingness to quit smoking.
* Do not read and understand Danish.
* Is not willing to cooperate with the clinic staff.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Active smokers who wish to quit
Sampling Method: Non-Probability Sample
Enrollment: 544 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Share of participants not smoking six months after the quit date. Intention-to-treat calculation, where participants lost to follow-up are included in as continued smokers | 6 months

SECONDARY OUTCOMES:
Share of participants not smoking six months after the quit date Per protocol calculation (participants lost to follow-up are excluded in the calculation of the quit rate) | 6 months
Share of participants at six months not smoking the last 14 days Intention-to-treat calculation, where participants lost to follow-up are included in as continued smokers | 6 months
Share of participants at six months not smoking the last 14 days Per protocol calculation (participants lost to follow-up are excluded in the calculation of the quit rate) | 6 months
Share of participants not smoking at the last visit at the GP Intention-to-treat calculation, where participants lost to follow-up are included in as continued smokers | 6 months
Share of participants not smoking at the last visit at the GP. Per protocol calculation (participants lost to follow-up are excluded in the calculation of the quit rate) | 6 months
Share of participants still smoking at six months with a reduction in the use of tobacco and the resulting reduction in smoking Intention-to-treat calculation, where participants lost to follow-up are included in as continued | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3051150&StudyName=Escape%20Smoke%20Project%3A%20Non-Intervention%20Non-Drug%20Multicenter%20Study%20on%20the%20Real-life%20Effectiveness%20of%20Smoking%20Cessation%20in%20General%20Practice%20